CLINICAL TRIAL: NCT07186322
Title: Fat Grafting in Upper Limb Burns Scars: a Randomized Clinical Trial
Brief Title: Autologous Fat Grafting in Upper Limb Burns Scars
Acronym: BURNSCARCARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Oliveira Mourão Junior, PHD Graduate in Translational Surgery. Plastic Surgery Division Resident, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7723619; U1111-1325-8730 (Other: Universal Trial Number - WHO)
Record Dates: First submitted 2025-08-06; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autologous Fat Grafting; Burn; Corticosteroid Injection
Keywords: randomized clinical trial; burns; autologous fat grafting; corticosteroid injection
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, single-center clinical trial with a parallel assignment design. Eligible adult patients with upper limb burn sequelae (functional contractures and/or pathological scars) will be randomly assigned in a 1:1 ratio to one of two treatment groups: (1) autologous fat grafting or (2) standard treatment (corticosteroid injection). Randomization will be conducted using a secure, computer-generated sequence through sealed opaque envelopes. Masking will be used only for the outcomes assessment; both patients and investigators will be aware of the assigned intervention. Participants will be followed for 6 months after treatment and evaluated at baseline and during follow-up using validated instruments. The primary objective is to compare the effectiveness of fat grafting versus standard treatment in improving scar quality and upper limb function.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. Although participants and treating physicians will be aware of the assigned intervention (open-label), outcome assessment will be blinded. At the 6-month follow-up, standardized clinical photographs of the treated areas will be obtained under controlled conditions and independently evaluated by an external assessor who will be blinded to the treatment group. This approach aims to minimize bias in the subjective assessment of scar quality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Fat Graft (Experimental): Participants randomized to this group will undergo autologous fat grafting to the affected areas of the upper limbs. The procedure includes harvesting adipose tissue via liposuction (typically from the abdomen or flanks), processing the fat through decantation and gentle emulsification, and reinjecting it into the burn sequelae areas using microcannulas in a layered, fanning technique. The intervention is performed in a single session under local or regional anesthesia depending on the case.
  Interventions: Procedure: Fat Graft
- Control Group - Corticosteroid Injection (Active Comparator): Participants in this group will receive standard care for burn scar sequelae, based on clinical judgment. This includes corticosteroid injections (triamcinolone 40 mg) for hypertrophic scars. The choice of intervention will follow standard clinical practice and will be documented in the protocol.
  Interventions: Procedure: Fat Graft

INTERVENTIONS:
Procedure: Fat Graft — Non-regenerative standard treatment for post-burn sequelae, involving either corticosteroid injection to reduce scar inflammation and fibrosis, or surgical release for contractures. The procedure type will be chosen based on the clinical indication and severity.

SUMMARY:
Burn injuries are a complex form of trauma with a high risk of complications. When they affect the upper limbs, patients often develop functional contractures and/or pathological scars that significantly impair mobility, quality of life, and psychological well-being. Current treatments-such as surgical interventions and corticosteroid injections-offer limited effectiveness, require prolonged therapy, and are associated with discomfort, multiple sessions, and indirect costs. Autologous fat grafting, a regenerative technique based on the transfer of the patient's own adipose tissue, has emerged as a promising alternative. It combines biocompatibility with regenerative and anti-inflammatory properties that may improve both function and scar quality. This randomized clinical trial aims to evaluate the efficacy of fat grafting in patients with post-burn upper limb sequelae compared to standard treatment (surgical release and/or corticosteroid injections). Patients will be prospectively followed and assessed using validated scar scales and functional outcomes.

DETAILED DESCRIPTION:
Burns represent a serious public health issue and are among the leading causes of trauma-related morbidity worldwide. Involvement of the upper limbs frequently results in long-term complications, including functional contractures and pathological scars, which compromise the patient's ability to return to daily activities and may severely affect quality of life. Traditionally, these sequelae are managed using surgical scar release procedures and/or corticosteroid injections. However, these conventional approaches have limitations: they provide only moderate efficacy, often require repeated sessions, and do not directly stimulate tissue regeneration. Furthermore, corticosteroid injections are associated with discomfort and risk of skin atrophy, and their repeated application can generate significant treatment fatigue.

Autologous fat grafting has gained attention in the context of regenerative medicine due to its dual ability to restore volume and promote cellular repair. The technique consists of harvesting adipose tissue from a donor area, processing it to concentrate regenerative elements (such as adipose-derived stem cells and growth factors), and injecting it into the target area. In the context of burn sequelae, fat grafting has demonstrated promising results in improving scar pliability, reducing pain and pruritus, and enhancing function, although high-quality randomized clinical trials remain scarce.

This study will enroll adult patients with a history of upper limb burns presenting with functional limitations and/or symptomatic pathological scars (e.g., hypertrophic scars, painful or pruritic areas). Participants will be randomly assigned to one of two treatment groups:

Experimental Group: Undergoing autologous fat grafting in the affected areas. Control Group: Receiving standard treatment, including corticosteroid injections and/or surgical scar release based on clinical indication.

Patients will be followed prospectively at predetermined time points and assessed using validated tools such as the Patient and Observer Scar Assessment Scale (POSAS), the Patient Scar Assessment Scale (PSAQ) and the Vancouver Scar Scale (VSS). Pain and pruritus intensity will be documented using visual analog scales (VAS). The study's primary endpoint will be the improvement in scar quality and function at 6 months. Secondary outcomes include patient satisfaction, pain reduction, cost-effectiveness, and the need for additional interventions.

The study complies with ethical standards, and all participants will provide informed consent. Given the limited availability of randomized trials in this field, the results of this study are expected to contribute robust scientific evidence to support or refute the use of fat grafting as a therapeutic modality for upper limb burn sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Presence of burn scars in the upper limbs (functional contractures and/or pathological scars)
* Scar area suitable for treatment (≥10 cm²)
* At least 12 months since the initial burn injury
* Willingness and ability to comply with study procedures and follow-up visits
* Signed informed consent form

Exclusion Criteria:

* Active local or systemic infection at the time of treatment
* Uncontrolled chronic diseases (e.g., diabetes mellitus with HbA1c > 8.0%)
* Use of systemic corticosteroids or immunosuppressants within 30 days before enrollment
* Previous surgical or injection treatment of the target scar within the past 6 months
* Known allergy to lidocaine or any material used in the procedures
* Coagulopathy or use of anticoagulant therapy
* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Scar Quality in Patient and Observer Scar Assessment Scale (POSAS) | 6 months after intervention
  The primary outcome is the change in scar quality in upper limb from baseline to 6 months post-treatment, as measured by a validated instruments:
  The Patient and Observer Scar Assessment Scale (POSAS), including both patient and observer domains (each scored 1-10, lower is better min: 6 points and maximum 60 points). Higher scores indicate worse scarring.

SECONDARY OUTCOMES:
Need for Additional Interventions | 6 month
  Number and type of additional procedures (e.g., re-injection, new surgical release, corticosteroid reapplication) required during the follow-up period.
Incidence of Adverse Events | 1 week, 1 month and 6 month
  Occurrence of treatment-related complications such as fat necrosis, infection, contour irregularities, delayed healing, or systemic adverse events.
Scar improvment measure by other scales - Patient Scar Assessment Scale | 6 month
  Measured in days from intervention to return to pre-injury activity level or occupational function. Reduction in pain and itching symptoms associated with burn scars, measured using and Patient Scar Assessment Scale (PSAQ). Scores vary depending on the version and domains used (e.g., appearance, symptoms, consciousness, satisfaction with appearance, satisfaction with symptoms). Each item is rated on a 4-point scale, and composite scores are calculated for each domain. Higher scores indicate worse patient-perceived scar quality and lower satisfaction.
Scar improvment measure by other scales - Vancouver Scar Scale | 6 month
  Measured in days from intervention to return to pre-injury activity level or occupational function Reduction in pain and itching symptoms associated with burn scars, measured using Vancouver Scar Scale (VSS). Total scores range from 0 to 13, based on four parameters (vascularity, pigmentation, pliability, and height). Lower scores indicate more normal scar characteristics; higher scores reflect worse scar severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University Of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study. Although the data will be de-identified, the nature of the study population and clinical context may still pose a residual risk of re-identification. Additionally, institutional policies and ethical considerations restrict public sharing of participant-level data without explicit consent for secondary use.

REFERENCES:
- [Result] Hoerst K, van den Broek L, Sachse C, Klein O, von Fritschen U, Gibbs S, Hedtrich S. Regenerative potential of adipocytes in hypertrophic scars is mediated by myofibroblast reprogramming. J Mol Med (Berl). 2019 Jun;97(6):761-775. doi: 10.1007/s00109-019-01772-2. Epub 2019 Mar 19. PMID 30891616
- [Result] Karakol P, Bozkurt M. Recent strategic approach in postburn extremity scars and contractures. J Plast Surg Hand Surg. 2021 Jun;55(3):153-161. doi: 10.1080/2000656X.2020.1856670. Epub 2020 Dec 14. PMID 33315507
- [Result] Jaspers MEH, Brouwer KM, van Trier AJM, Middelkoop E, van Zuijlen PPM. Sustainable effectiveness of single-treatment autologous fat grafting in adherent scars. Wound Repair Regen. 2017 Apr;25(2):316-319. doi: 10.1111/wrr.12521. Epub 2017 Apr 24. PMID 28370844
- [Result] Simonacci F, Bertozzi N, Grieco MP, Grignaffini E, Raposio E. Procedure, applications, and outcomes of autologous fat grafting. Ann Med Surg (Lond). 2017 Jun 27;20:49-60. doi: 10.1016/j.amsu.2017.06.059. eCollection 2017 Aug. PMID 28702187
- [Result] Negenborn VL, Groen JW, Smit JM, Niessen FB, Mullender MG. The Use of Autologous Fat Grafting for Treatment of Scar Tissue and Scar-Related Conditions: A Systematic Review. Plast Reconstr Surg. 2016 Jan;137(1):31e-43e. doi: 10.1097/PRS.0000000000001850. PMID 26710059
- [Result] Jaspers MEH, Brouwer KM, Middelkoop E, van Zuijlen PPM. Autologous fat grafting; it almost seems too good to be true. Burns. 2017 May;43(3):690-691. doi: 10.1016/j.burns.2017.01.039. Epub 2017 Mar 1. No abstract available. PMID 28258778
- [Result] Lesmanawati FE, Windura CA, Saputro ID, Hariani L. Autologous fat grafting and adipose-derived stem cells therapy for acute burns and burn-related scar: A systematic review. Tzu Chi Med J. 2024 Mar 6;36(2):203-211. doi: 10.4103/tcmj.tcmj_189_23. eCollection 2024 Apr-Jun. PMID 38645780
- [Result] Abu Alqam R, Alshammari AJ, Alkhwildi LA, Bamatraf MS, Khashab RM, Al Dwehji AMO, Alsuayri RA, Fadel ZT. Effectiveness of Autologous Fat Grafting in the Treatment of Scars: A Systematic Review and Meta-Analysis. Aesthetic Plast Surg. 2024 Oct;48(19):3945-3961. doi: 10.1007/s00266-024-04131-w. Epub 2024 Jul 16. PMID 39014237
- [Result] Piccolo NS, Piccolo MS, Piccolo MT. Fat grafting for treatment of burns, burn scars, and other difficult wounds. Clin Plast Surg. 2015 Apr;42(2):263-83. doi: 10.1016/j.cps.2014.12.009. Epub 2015 Feb 21. PMID 25827568
- [Result] Durani P, McGrouther DA, Ferguson MW. The Patient Scar Assessment Questionnaire: a reliable and valid patient-reported outcomes measure for linear scars. Plast Reconstr Surg. 2009 May;123(5):1481-1489. doi: 10.1097/PRS.0b013e3181a205de. PMID 19407619
- [Result] 28. Linhares CB, Viaro MSS, Collares MVM et al. Tradução para o português da Patient and Observer Scar Assessment Scale (POSAS). Rev Bras Cir Plást. 2016;31(1):95-100.
- [Result] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Result] 26. Santos MC, Tibola J, Marques CMG. Tradução, revalidação e confiabilidade da Escala de Cicatrização de Vancouver para língua portuguesa - Brasil. Rev Bras Queimaduras. 2014;13(1):26-3.
- [Result] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Result] Spiekman M, Przybyt E, Plantinga JA, Gibbs S, van der Lei B, Harmsen MC. Adipose tissue-derived stromal cells inhibit TGF-beta1-induced differentiation of human dermal fibroblasts and keloid scar-derived fibroblasts in a paracrine fashion. Plast Reconstr Surg. 2014 Oct;134(4):699-712. doi: 10.1097/PRS.0000000000000504. PMID 25357030
- [Result] Hong SJ, Traktuev DO, March KL. Therapeutic potential of adipose-derived stem cells in vascular growth and tissue repair. Curr Opin Organ Transplant. 2010 Feb;15(1):86-91. doi: 10.1097/MOT.0b013e328334f074. PMID 19949335
- [Result] Tan SS, Ng ZY, Zhan W, Rozen W. Role of Adipose-derived Stem Cells in Fat Grafting and Reconstructive Surgery. J Cutan Aesthet Surg. 2016 Jul-Sep;9(3):152-156. doi: 10.4103/0974-2077.191672. PMID 27761084
- [Result] Gir P, Brown SA, Oni G, Kashefi N, Mojallal A, Rohrich RJ. Fat grafting: evidence-based review on autologous fat harvesting, processing, reinjection, and storage. Plast Reconstr Surg. 2012 Jul;130(1):249-258. doi: 10.1097/PRS.0b013e318254b4d3. PMID 22743888
- [Result] Gutowski KA; ASPS Fat Graft Task Force. Current applications and safety of autologous fat grafts: a report of the ASPS fat graft task force. Plast Reconstr Surg. 2009 Jul;124(1):272-280. doi: 10.1097/PRS.0b013e3181a09506. PMID 19346997
- [Result] 18. Poon R, Messa CA, Moquin A, et al. Complications associated with autologous fat grafting: A systematic review. Aesthet Surg J. 2021;41(9):NP1336-NP1348.
- [Result] 17. Schroeder A, Pinheiro LHZ, Angeline JR, et al. Análise de complicações de lipoenxertias realizadas em hospital público universitário entre 2015 e 2018: Estudo retrospectivo transversal. Rev Bras Cir Plást. 2022.
- [Result] Rigotti G, Marchi A, Galie M, Baroni G, Benati D, Krampera M, Pasini A, Sbarbati A. Clinical treatment of radiotherapy tissue damage by lipoaspirate transplant: a healing process mediated by adipose-derived adult stem cells. Plast Reconstr Surg. 2007 Apr 15;119(5):1409-1422. doi: 10.1097/01.prs.0000256047.47909.71. PMID 17415234
- [Result] 14. Rammelt S, Zwipp H. Lipoaspirate transfer for the treatment of posttraumatic and postburn soft tissue defects. Eur J Trauma Emerg Surg. 2015;41(3):277-285.
- [Result] Klinger M, Caviggioli F, Klinger FM, Giannasi S, Bandi V, Banzatti B, Forcellini D, Maione L, Catania B, Vinci V. Autologous fat graft in scar treatment. J Craniofac Surg. 2013 Sep;24(5):1610-5. doi: 10.1097/SCS.0b013e3182a24548. PMID 24036737
- [Result] Pierini É, Assunção FF de O. Aesthetic resources applied to burns: literature review. Manual Therapy, Posturology & Rehabilitation Journal
- [Result] 11. Moreira JM, Braga NCC, Abrahao A, et al. Associação da lipoenxertia no tratamento de cicatrizes de queimadura: Um relato de caso. BJD. 2020;6(11):93200-93211
- [Result] 10. Popp D, Branski LK, Kamolz LP. Long-Term Sequelae of Burn Injury: Current Understanding of Pathophysiology, Therapeutic, and Rehabilitative Options with an Emphasis on Hypertrophic Scarring and Laser Therapy
- [Result] Xie C, Hu J, Cheng Y, Yao Z. Researches on cognitive sequelae of burn injury: Current status and advances. Front Neurosci. 2022 Nov 4;16:1026152. doi: 10.3389/fnins.2022.1026152. eCollection 2022. PMID 36408414
- [Result] 7. Caldas YC, Souza IML, Souza KL, Gazé LA, Baia VRV, Monteiro RPA. Avaliação do desempenho ocupacional de paciente queimado pós-alta hospitalar. Rev Interinstit Bras Ter Ocup. 2019.
- [Result] 5. WORLD HEALTH ORGANIZATION. A WHO plan for burn prevention and care. Geneva: WHO, 2008. Disponível em: https://apps.who.int/iris/bitstream/handle/10665/97852/9789241596299_eng.pdf. Acesso em: 11 jan. 2025.
- [Result] 4. American Burn Association. National Burn Repository 2019 Update. Report of Data from 2008-2018. Available online: https://sk75w2kudjd3fv2xs2cvymrgwpengine.netdna- ssl.com/wpcontent/uploads/2020/05/2019-ABA-Annual-Report_FINAL.pdf.
- [Result] Gibson JAG, Yarrow J, Brown L, Evans J, Rogers SN, Spencer S, Shokrollahi K. Identifying patient concerns during consultations in tertiary burns services: development of the Adult Burns Patient Concerns Inventory. BMJ Open. 2019 Dec 30;9(12):e032785. doi: 10.1136/bmjopen-2019-032785. PMID 31892660
- [Result] Al Ghriwati N, Sutter M, Pierce BS, Perrin PB, Wiechman SA, Schneider JC. Two-Year Gender Differences in Satisfaction With Appearance After Burn Injury and Prediction of Five-Year Depression: A Latent Growth Curve Approach. Arch Phys Med Rehabil. 2017 Nov;98(11):2274-2279. doi: 10.1016/j.apmr.2017.04.011. Epub 2017 May 5. PMID 28483656
- [Result] Deeter L, Seaton M, Carrougher GJ, McMullen K, Mandell SP, Amtmann D, Gibran NS. Hospital-acquired complications alter quality of life in adult burn survivors: Report from a burn model system. Burns. 2019 Feb;45(1):42-47. doi: 10.1016/j.burns.2018.10.010. Epub 2018 Nov 23. PMID 30477817

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT07186322/Prot_SAP_000.pdf
  • Study Protocol and Informed Consent Form (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT07186322/Prot_ICF_001.pdf